CLINICAL TRIAL: NCT03118778
Title: Proton Pump Inhibitor (PPI) Inappropriate Use and Economic Burden in Chinese Population: A Descriptive Retrospective Observational Study Using Database
Brief Title: Proton Pump Inhibitor (PPI) Inappropriate Use and Economic Burden in Chinese Population
Acronym: ECHO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9612R00010
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Gastrointestinal Disease
Keywords: Stress Ulcer Prevention
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive retrospective database analysis study in using database. All patients with a physician PPI prescription will be selected to estimate the PPI inappropriate use.

DETAILED DESCRIPTION:
Study primary objective is to identify the inappropriate use of PPI (overall, outpatient & inpatient).

ELIGIBILITY:
Inclusion Criteria:

* All patients in 2015 China Health Insurance Research Association (CHIRA) database.
* Patients had PPI prescription during Jan. 2015 to Dec. 2015 will be selected to estimate the PPI inappropriate use.

Exclusion Criteria:

• Patients without data of treatment information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were prescribed PPIs during Jan. 2015 to Dec. 2015 will be identified and then all their inpatient and outpatient information will be extracted.
Sampling Method: Non-Probability Sample
Enrollment: 90895 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Overall proportion of patient inappropriate use of PPI | 2015.01-2015.12
  Overall number of patient times/courses with PPI inappropriate use (including non-indication use, over maximum daily dose and over maximum duration) divided by the total number of patient-times/courses with PPI use for both outpatients and inpatients.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: D9612R00010_CSR-Synopsis_V 1.0-20180629 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14674&filename=D9612R00010_CSR-Synopsis_V%201.0-20180629.pdf